CLINICAL TRIAL: NCT05369312
Title: Phase 1 Study of BPI-442096 in Advanced Solid Tumor Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BTP-661711
Record Dates: First submitted 2022-05-05; First posted 2022-05-11 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-04

CONDITIONS: Solid Tumor; Non-small Cell Lung Cancer; Pancreatic Cancer; Colorectal Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Oral tablets taken in escalating levels to determine MTD/RP2D. Each treatment cycle will be 21 days in duration with BPI-442096 administered, once daily (QD).
  Interventions: Drug: BPI-442096
- Dose Expansion (Experimental): Oral tablets administered at MTD/RP2D defined dose. Each treatment cycle will be 21 days in duration with BPI-442096 administered, once daily (QD)
  Interventions: Drug: BPI-442096

INTERVENTIONS:
Drug: BPI-442096 — Subjects will receive BPI-442096 until disease progression

SUMMARY:
A first-in-human study to evaluate the safety, tolerability and maximum tolerated dose (MTD) and establish the recommended phase 2 dose (RP2D) of BPI-442096, a SHP2 inhibitor, in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The first-in-human (FIH) study of BPI-442096 will be an open-label, non-randomized, Phase 1 study utilizing a modified "3+3" dose escalation followed by an expansion phase in patients with KRAS G12 mutation, class-3 BRAF mutation, NF1 LOF mutation or RTK mutation, amplification or rearrangement advanced solid tumors. The primary objective is to determine safety and tolerability of BPI-442096, the MTD and RP2D. The secondary objectives are to assess the pharmacokinetic (PK) and pharmacodynamic (PD) profile, preliminary anti-tumor activity of BPI-442096.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Age ≥18 and ≤75 years, male and female patients;
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1;
* Dose escalation phase: histologically or cytologically confirmed locally advanced or metastatic solid tumor patients (excluding HCC patients), who had disease progression after standard therapy, intolerable to standard therapy, refuse to standard therapy or for whom no standard therapy exists;
* Dose expansion phase: histologically or cytologically confirmed locally advanced non-small cell lung cancer, pancreatic cancer, colorectal cancer or other diagnosed solid tumor patients (excluding HCC patients), who had disease progression after standard therapy, intolerable to standard therapy, refuse to standard therapy or for whom no standard therapy exists;
* Evaluable lesion required for dose escalation phase and at least 1 measurable lesion as per RECIST v1.1 required for dose expansion phase;
* Dose expansion only: Patients must have confirmation of tumour mutation status (including KRAS G12, Class-3 BRAF, NF1 LOF mutations, RTK mutations, amplifications or rearrangements).
* Adequate organ function;

Exclusion Criteria:

* Patients who have previously received a SHP2 inhibitor;
* Inadequate wash-out of prior therapies described per protocol, which may include anti-tumor therapies, tumor adjuvant drugs, organ or stem cell transplantation, moderate or strong CYP3A inhibitor or inducer;
* Patients with severe or unstable systemic disease, unstable/symptomatic CNS metastasis, other malignant tumors, autoimmune disease, ILD, cardiac disease, bleeding or embolic disease, infectious disease, conditions affecting drug swallow and absorption, medical history leading to chronic diarrhea, etc;
* Pregnancy or lactation;
* Other conditions considered not appropriate to participate in this trial by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
The adverse events (AEs) | Through the Phase I, approximately 24 months
  Safety and tolerability will be assessed by monitoring frequency, duration and severity of adverse events (AEs).
Determine the recommended Phase II dose (RP2D) | Through the Phase I, approximately 24 months
  Number of subjects with dose limiting toxicity

SECONDARY OUTCOMES:
Cmax | Through the Phase I, approximately 24 months
  Maximum observed concentration
Tmax | Through the Phase I, approximately 24 months
  Time to reach maximum observed plasma concentration
t1/2 | Through the Phase I, approximately 24 months
  Half-life time
AUC0-t | Through the Phase I, approximately 24 months
  Area under the concentration-time curve from time 0 to t
the objective response rate (ORR） | Through the Phase I, approximately 24 months
  The proportion of patients with complete response (CR) and partial response (PR) in all patients
Disease control rate (DCR） | Through the Phase I, approximately 24 months
  The proportion of patients with CR, PR and stable disease (SD) in all patients
Duration of response (DOR） | Through the Phase I, approximately 24 months
  The time from the first CR or PR to the first PD or death due to any cause
Progression free survival (PFS) | Through the Phase I, approximately 24 months
  The time from the date of randomization to disease progression (PD) or death, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, Ph.D, Principal Investigator — Guangdong Provincial People's Hospital
Locations (5):
- China (5):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun yat-sen university, Guangzhou, Guangdong
  - Henan Tumor Hospital, Zhengzhou, Henan
  - Zhongshan Hospital affiliated to Fudan University, Xuhui, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No